CLINICAL TRIAL: NCT06715046
Title: Cell Free DNA Profiling As a Tool to Monitor Clinically-Relevant Events in Allogeneic Hematopoietic Stem Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: University of Turin, Italy (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvia Deaglio, Professor of Medical Genetics, University of Turin, Italy
Other Study IDs: P2022ZRF5H
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: GVHD - Graft-Versus-Host Disease; Infections After HSCT; Transplant Associated Microangiopathy TAM; Sinusoidal Obstruction Syndrome (SOS); HSCT Engraftment
Keywords: cfDNA; methylation; epigenetic profile; HSCT; liquid biopsy
MeSH Terms: conditions — Graft vs Host Disease; Hepatic Veno-Occlusive Disease | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will undergo cfDNA extraction. Resulting sample will be analyzed for the purposes of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- GVHD patients: This group gathers all the patients that eventually develop GVHD
  Interventions: Diagnostic Test: Sample collation for cfDNA methylation analysis; Diagnostic Test: Sample collection for EV phenotype analysis
- Control patients: This group gathers all the patients that will not develop post-HSCT complications and show no signs of relapse.
  Interventions: Diagnostic Test: Sample collation for cfDNA methylation analysis; Diagnostic Test: Sample collection for EV phenotype analysis
- Infection patients: This group gathers all the patients that develop post-HSCT infections
  Interventions: Diagnostic Test: Sample collation for cfDNA methylation analysis; Diagnostic Test: Sample collection for EV phenotype analysis
- Relapse patients: This group gathers all the patients that relapse after HSCT
  Interventions: Diagnostic Test: Sample collation for cfDNA methylation analysis; Diagnostic Test: Sample collection for EV phenotype analysis
- TAD/SOS patients: This goup gathers patients presenting with transplant associated microangiopathy or sinusoidal obstruction.

INTERVENTIONS:
Diagnostic Test: Sample collation for cfDNA methylation analysis — Sample collation for cfDNA methylation analysis
  Groups: Control patients; GVHD patients; Infection patients; Relapse patients
Diagnostic Test: Sample collection for EV phenotype analysis — Analysis of the EV phenotype to evaluate their potential value as markers for GVHD, relapse and engraftment.
  Groups: Control patients; GVHD patients; Infection patients; Relapse patients

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (HSCT) is a life-saving treatment for people with severe blood-related diseases. However, it comes with serious risks, including a condition called graft-versus-host disease (GVHD), where the transplanted cells attack the patient's body. GVHD can occur in about 50% of patients acutely and 35% in a chronic form, potentially affecting organs like the skin, liver, and gastrointestinal system. Currently, doctors diagnose GVHD based on symptoms, as there are no easy tests available.

Infections can also be a problem after HSCT, as dormant viruses may reactivate. These infections are monitored using specialized tests. Additionally, doctors use advanced methods, like analyzing minimal residual disease (MRD) and chimerism, to check for the risk of the original disease coming back. MRD is tracked by looking for specific genetic markers of the disease in the patient's blood or bone marrow.

Another emerging tool involves analyzing cell-free DNA (cfDNA)-tiny fragments of DNA found in bodily fluids that come from dying cells. This technique, called liquid biopsy, has been revolutionary in areas like cancer detection, pregnancy testing, and organ transplants. For example, in organ transplants, cfDNA can indicate early signs of rejection, helping reduce the need for invasive biopsies.

In HSCT, the use of cfDNA to monitor complications like GVHD or relapse has not been fully explored. This pilot study aims to investigate whether analyzing cfDNA using a technique called epigenomic profiling can help detect acute GVHD, as well as other post-transplant issues like infections, disease relapse, and chronic GVHD. The goal is to compare cfDNA analysis to current testing methods to see if it offers better or earlier detection of complications.

This research could pave the way for improved, less invasive monitoring of HSCT patients, potentially leading to better outcomes and fewer complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be affected by an hematological malignancy requiring hematopoietic stem cell transplantation (HSCT).

Exclusion Criteria:

* Patients can not be 17 years old or yunger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled at the Unità di Ematologia e Trapianto di Midollo Osseo e Oncoematologia of the San Raffaele Hospital in Milan and at the SS Trapianto allogenico e terapie cellulari, SC Ematologia U of the Città della Salute e della Scienza Hospital in Turin.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Epigenetic profiling of cfDNA in patients developing GVHD | From enrollment to the end of post-HSCT follow-up of 12 months
  Analysis of cfDNA methylation patterns in GVHD patients vs controls to define potential marker regions to be translationally utilized for early detections of the disease.

SECONDARY OUTCOMES:
Epigenetic profiling of cfDNA in patients developing post-HSCT infections | From enrollment to the end of post-HSCT follow-up of 12 months
  Analysis of cfDNA methylation patterns in patients developing post-HSCT transplantation infections vs controls to define potential marker regions to be translationally utilized for early detections of the condition.
Epigenetic profiling of cfDNA in patients with engraftment failure | From enrollment to the end of post-HSCT follow-up of 12 months
  Analysis of cfDNA methylation patterns in patients with engraftment failure vs controls.
Epigenetic profiling of cfDNA in relapsing patients | From enrollment to the end of post-HSCT follow-up of 12 months
  Description: Analysis of cfDNA methylation patterns in relapsing patients vs controls.
Epigenetic profiling of cfDNA in patients developing transplant associated microangiopathy or sinusoidal obstruction | From enrollment to the end of post-HSCT follow-up of 12 months
Evaluation of EV phenotype | From enrollment to the end of post-HSCT follow-up of 12 months
  Evaluation of circulating vesicle phenotype in as potential biomarker for GVHD, engraftment and relapse.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Unità di Ematologia e Trapianto di Midollo Osseo e Oncoematologia of the San Raffaele Hospital in Milan, Milan, Milan
  - SS Trapianto allogenico e terapie cellulari, SC Ematologia U of the Città della Salute e della Scienza Hospital, Turin, Turin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang X, He B. Insight into endothelial cell-derived extracellular vesicles in cardiovascular disease: Molecular mechanisms and clinical implications. Pharmacol Res. 2024 Sep;207:107309. doi: 10.1016/j.phrs.2024.107309. Epub 2024 Jul 14. PMID 39009292
- [Background] Jodele S, Dandoy CE, Sabulski A, Koo J, Lane A, Myers KC, Wallace G, Chima RS, Teusink-Cross A, Hirsch R, Ryan TD, Benoit S, Davies SM. Transplantation-Associated Thrombotic Microangiopathy Risk Stratification: Is There a Window of Opportunity to Improve Outcomes? Transplant Cell Ther. 2022 Jul;28(7):392.e1-392.e9. doi: 10.1016/j.jtct.2022.04.019. Epub 2022 Apr 29. PMID 35490975
- [Background] Avni B, Neiman D, Shaked E, Gal-Rosenberg O, Grisariu S, Kuzli M, Avni I, Fracchia A, Stepensky P, Zuckerman T, Lev-Sagie A, Fox-Fisher I, Piyanzin S, Moss J, Salpeter SJ, Glaser B, Shemer R, Dor Y. Chronic graft-versus-host disease detected by tissue-specific cell-free DNA methylation biomarkers. J Clin Invest. 2024 Jan 16;134(2):e163541. doi: 10.1172/JCI163541. PMID 37971879
- [Background] Oellerich M, Budde K, Osmanodja B, Bornemann-Kolatzki K, Beck J, Schutz E, Walson PD. Donor-derived cell-free DNA as a diagnostic tool in transplantation. Front Genet. 2022 Oct 21;13:1031894. doi: 10.3389/fgene.2022.1031894. eCollection 2022. PMID 36339004
- [Background] Cheng AP, Cheng MP, Loy CJ, Lenz JS, Chen K, Smalling S, Burnham P, Timblin KM, Orejas JL, Silverman E, Polak P, Marty FM, Ritz J, De Vlaminck I. Cell-free DNA profiling informs all major complications of hematopoietic cell transplantation. Proc Natl Acad Sci U S A. 2022 Jan 25;119(4):e2113476118. doi: 10.1073/pnas.2113476118. PMID 35058359